CLINICAL TRIAL: NCT00014274
Title: Randomized Phase II/III Study Assessing Gemcitabine/Carboplatin And Methotrexate/Carboplatin/Vinblastine In Previously Untreated Patients With Advanced Urothelial Cancer Ineligible For Cisplatin Based Chemotherapy
Brief Title: Combination Chemotherapy in Treating Patients With Transitional Cell Cancer of the Urothelium
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30986; EORTC-GU-30986
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Gemcitabine; Methotrexate; Vinblastine

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: methotrexate
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective for transitional cell cancer of the urothelium.

PURPOSE: Randomized phase II/III trial to compare different combination chemotherapy regimens in treating patients who have transitional cell cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the antitumor activity of gemcitabine and carboplatin vs methotrexate, carboplatin, and vinblastine in patients with transitional cell cancer of the urothelium who are ineligible for cisplatin-based chemotherapy.
* Compare the toxicity and acute and intermediate (1-2 years) side effects of these regimens in these patients.
* Compare the complete response rates, progression-free survival, and overall survival of patients treated with these regimens.
* Compare the symptoms and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive methotrexate* IV and vinblastine IV on days 1, 15, and 22 and carboplatin IV over 1 hour on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: * Methotrexate is omitted for patients with pleural effusion or ascites until complete resolution and for patients with a glomerular filtration rate less than 30 mL/min or creatinine greater than 2 mg/dL

Patients in either arm who achieve a complete response (CR) receive 2 additional courses of chemotherapy beyond CR.

Quality of life is assessed at baseline, after every 2 courses of chemotherapy, and within 6 weeks of completion of therapy.

Patients are followed within 6 weeks, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 156 patients (78 per treatment arm) will be accrued for the phase II portion of this study. A total of 225 patients will be accrued for the phase II + III portions of this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell cancer of the urothelium, including the renal pelvis, ureters, urinary bladder, and urethra, meeting 1 of the following criteria:

  * Unresected positive lymph node
  * Distant metastases (M1, stage IV)
  * Unresectable primary bladder cancer (T3-4)
* Measurable disease
* Ineligible for cisplatin-based chemotherapy and presenting with the following:

  * WHO performance status 2 AND/OR
  * Glomerular filtration rate greater than 30 mL/min but less than 60 mL/min
* No brain metastases or other CNS lesions

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 125,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times normal
* AST/ALT no greater than 3 times normal (5 times normal if liver metastases are present)

Renal:

* See Disease Characteristics
* Calcium normal

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study participation
* No psychological, familial, sociological, or geographical condition that would preclude study participation
* No other prior or concurrent malignancy except cured basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior systemic biologic therapy

Chemotherapy:

* See Disease Characteristics
* No prior systemic cytotoxic therapy (including adjuvant and neoadjuvant chemotherapy)

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 months since prior radiotherapy
* Prior radiotherapy to study lesions allowed if there is evidence of disease progression

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2001-01; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Duration of survival

SECONDARY OUTCOMES:
Response as assessed by RECIST criteria
Toxicity as assessed by CTC v2

CONTACTS AND LOCATIONS:
Overall Officials: Gerwin Kaiser, MD, Study Chair — Klinikum Nuernberg - Klinikum Nord
Locations (29):
- Austria (2):
  - St. Johanns-Spital, Salzburg
  - Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Groeninge - Oncologisch Centrum, Kortrijk
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Klinikum Nuernberg - Klinikum Nord, Nuremberg, Germany
- National Institute of Oncology, Budapest, Hungary
- Assaf Harofeh Medical Center, Ẕerifin, Israel
- Italy (2):
  - Universita Di Palermo, Palermo
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Spain (5):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Instituto Valenciano De Oncologia, Valencia
- United Kingdom (4):
  - Leeds Cancer Centre at St. James's University Hospital, Southampton, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England

REFERENCES:
- [Result] De Santis M, Bellmunt J, Mead G, Kerst JM, Leahy M, Maroto P, Gil T, Marreaud S, Daugaard G, Skoneczna I, Collette S, Lorent J, de Wit R, Sylvester R. Randomized phase II/III trial assessing gemcitabine/carboplatin and methotrexate/carboplatin/vinblastine in patients with advanced urothelial cancer who are unfit for cisplatin-based chemotherapy: EORTC study 30986. J Clin Oncol. 2012 Jan 10;30(2):191-9. doi: 10.1200/JCO.2011.37.3571. Epub 2011 Dec 12. PMID 22162575
- [Result] De Santis M, Bellmunt J, Mead G, Kerst JM, Leahy M, Maroto P, Skoneczna I, Marreaud S, de Wit R, Sylvester R. Randomized phase II/III trial assessing gemcitabine/ carboplatin and methotrexate/carboplatin/vinblastine in patients with advanced urothelial cancer "unfit" for cisplatin-based chemotherapy: phase II--results of EORTC study 30986. J Clin Oncol. 2009 Nov 20;27(33):5634-9. doi: 10.1200/JCO.2008.21.4924. Epub 2009 Sep 28. PMID 19786668
- [Result] De Santis M, Bellmunt J, Mead B, et al.: Randomized phase II/III study assessing gemcitabine/carboplatin (GC) and methotrexate/carboplatin/vinblastine (M-CAVI) in previously untreated patients (pts) with advanced urothelial cancer ineligible for cisplatin based chemotherapy: phase II results of. [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-288, 2008.